CLINICAL TRIAL: NCT07359742
Title: Assessing Signatures for Fibrosis Detection in Chronic Liver Disease: A Step Beyond Conventional Biomarkers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CoMis Fib
Record Dates: First submitted 2025-12-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Chronic Liver Disease (CLD); Fibrosis of Liver
Keywords: chronic liver disease; fibrosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Blood Specimen Collection; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDTA tube (Experimental)
  Interventions: Other: Blood draw for biomarkers

INTERVENTIONS:
Other: Blood draw for biomarkers — EDTA tube Blood draw for biomarkers

SUMMARY:
Morbidity and mortality of CLD is driven by the extent of liver fibrosis, characterized by scar formation and disruption of the normal liver architecture. HSCs play a central role in liver fibrosis development. When hepatocytes are damaged, HSCs undergo myofibroblast differentiation, transitioning into an activated state. So far, no efficient biomarkers can estimate the degree of HSC activation or reversal across all aetiologies of CLD, although this could be a more sensitive marker than fibrosis measurement which is secondary to HSC activation. This study aims to correlate biomarkers to the fibrosis stage in a larger cohort of patients with CLD across all aetiologies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18y
* Chronic liver disease: alcohol, metabolic dysfunction associated steatotic liver disease, viral hepatitis, autoimmune hepatitis, cholestatic liver disease and hemochromatosis

Exclusion Criteria:

* <18y
* Acute hepatitis
* Contra-indication for transient elastography (Fibroscan®) such as ascites or overt heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
correlation of biomarkers in blood and fibrosis stage of liver | Day 1 of the study
  correlation of biomarkers in blood and fibrosis stage of the liver (comparison with: transient elastography, fib4, APRI and liver biopsy if possible)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No